CLINICAL TRIAL: NCT03583203
Title: Efficacy in Patients With Severe Mental Disorders of an Intensive Motivational Interventional Programme Offering Individualized Information on Respiratory Damage for Smoking Cessation
Brief Title: Tobacco Intensive Motivational and Estimate Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Fernando Sarramea Crespo, Principal Investigator, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI16/0082
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Severe Mental Disorder; Smoking Cessation; COPD
Keywords: schizophrenia; bipolar disorder; tobacco; COPD
MeSH Terms: conditions — Mental Disorders; Smoking Cessation; Pulmonary Disease, Chronic Obstructive; Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will include personalized information about lung damage. After evaluating their COPD, the patients will be informed about its existence it so and staging. Depending on the damage found, the generation of motivation will focus on the different prevention methods. Likewise, after the motivation level is set, the patients will be offered the option of treatment and regular follow-up. The intervention will be strengthened by motivational messages, half of which are linked to the possibilities of preventing respiratory damage, sent to the patient's mobile phone via SMS during the 3 months after the face-to-face intervention. Patients without mobile phones will receive a call on their phone to convey the same messages.
  Interventions: Device: personalized information about lung damage
- Control Group (No Intervention): The control intervention lasts 30 minutes and will be structured around the 5 A's technique (Ask, Advice, Assess, Assist and Arrange).

INTERVENTIONS:
Device: personalized information about lung damage — Chronic obstructive pulmonary disease (COPD) will be evaluated using spirometry. Based on this value, a motivational message about prevention will be issued for the intervention group, which will be reinforced by individualized text messages over a period of 3 months
  Arms: Experimental Group

SUMMARY:
Randomized, open label, prospective study with a 12-month follow-up period. The primary objective evaluates the effectiveness of an intensive anti-smoking programme that informs patients of their individual risk of lung damages and the possibilities of prevention. The main measurement will be having given up smoking in month 12, measurement of self-reported abstinence on the 7 previous days and confirmed by a CO-oximeter test< 10 ppm, between the intervention and control group. A total of 9 urban and rural mental health centres will participate in the study. The intervention group will undergo spirometry and presence and the degree of respiratory obstruction will be assessed. Participants will be given individual information to generate a motivational message about the possibilities of prevention and the information will be maintained for three months by sending text messages (SMS) to their mobile phones. The efficacy of the method and the pulmonary damage variables will be evaluated: smoking cessation at the end of follow-up will be confirmed by cooximetry, and the COPD diagnosis and the severity of the staging for disease will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40 and 70
* Confirmed diagnosis of Bipolar Disorder or Schizophrenia according to Diagnostic and Statistical Manual of Mental Disorder IV (DSM-IV-TR)
* Active smokers who currently consume at least 10 cigarettes a day, with a cumulative consumption of 10 packets/year or more.

Exclusion Criteria:

* Previous respiratory diagnosis of: asthma, cystic fibrosis, tuberculosis, simple chronic bronchitis, restrictive pulmonary disease or bronchiectasis
* Acute respiratory symptoms
* Heart disease or advanced oncological processes
* Existence of a pathology which makes it advisable not to perform spirometry (recent pneumothorax, recent thoracic or abdominal surgery, aortic aneurysm, unstable angulation, retinal detachment, facial hemiparesis or oral/dental problems)
* Patients who, due to their intellectual disability or mental pathology, do not understand or cannot be forced to perform spirometry
* Clinical instability with results of over 14 points on the Hamilton Depression Rating Scale (HDRS), a Young Mania Rating Scale (YMRS) of over 6 or a Positive and Negative Syndrome Scale (PANSS) of over 70

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 12 months
  Self-reported abstinence over the previous 7 days, confirmed by cooximetry with expired CO <10 ppm
COPD diagnosis | 12 month
  Presence of COPD and staging and percentage of forced expiratory volume at one second (FEV1) compared with expected level

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Sarramea Crespo, Phd, Principal Investigator — Hospital Universitario Reina Sofia Cordoba
Locations (1):
- Fernando Sarramea Crespo, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jaen-Moreno MJ, Feu N, Redondo-Ecija J, Montiel FJ, Gomez C, Del Pozo GI, Alcala JA, Gutierrez-Rojas L, Balanza-Martinez V, Chauca GM, Carrion L, Osuna MI, Sanchez MD, Caro I, Ayora M, Valdivia F, Lopez MS, Poyato JM, Sarramea F. Smoking cessation opportunities in severe mental illness (tobacco intensive motivational and estimate risk - TIMER-): study protocol for a randomized controlled trial. Trials. 2019 Jan 14;20(1):47. doi: 10.1186/s13063-018-3139-9. PMID 30642365